CLINICAL TRIAL: NCT06074718
Title: Exploring the Therapeutic Effect of Pricking Therapy Combined With Wheat Grain Moxibustion on Malignant Tumors of Spleen Deficiency and Dampness Resistance Type
Brief Title: Clinical Value of Prick Therapy Combined With Wheat Grain Moxibustion in the Treatment of Spleen Deficiency and Dampness Obstructed Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Principal Investigator, niqingtao, Deputy Director, Project Management Department, Centre for Clinical Research, Jiangsu Taizhou People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JiangsuTaizhouPH
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pricking Therapy on the Back Shu Points; Wheat Grain Moxibustion on the Back Shu Points
Keywords: spleen deficiency and dampness obstructed; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pricking therapy and wheat grain moxibustion combined with chemotherapy (Experimental): pricking therapy and wheat grain moxibustion on the back shu points or positive reaction points combined with chemotherapy
  Interventions: Other: pricking therapy and wheat grain moxibustion
- chemotherapy (Active Comparator): Conventional chemotherapy regimen
  Interventions: Other: pricking therapy and wheat grain moxibustion

INTERVENTIONS:
Other: pricking therapy and wheat grain moxibustion — pricking therapy and wheat grain moxibustion on the back shu points or positive reaction points

SUMMARY:
This study aims to investigate the clinical efficacy and associated immune and inflammatory mechanisms in patients with malignant tumors of spleen deficiency and dampness resistance type, by applying pricking therapy and wheat grain moxibustion on the back shu points or positive reaction points.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Western medicine and traditional Chinese medicine for malignant tumors;
* Clinical diagnosis of spleen deficiency dampness obstruction in traditional Chinese medicine;
* Good compliance and signed informed consent form.

Exclusion Criteria:

* Patients who cannot lie prone for a long time;
* Pregnant women;
* Lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (ORR) | 3 years
  Evaluate the objective response rate (ORR) of subjects based on RECIST V1.1

SECONDARY OUTCOMES:
progression free survival (PFS), | 5 years
  Evaluate subjects' progression free survival (PFS), overall survival (OS), and duration of remission (DOR) based on RECIST V1.1
overall survival (OS) | 5 years
  Evaluate subjects' overall survival (OS) based on RECIST V1.1
duration of remission (DOR) | 5 years
  Evaluate subjects' duration of remission (DOR) based on RECIST V1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Qingtao Ni, Taizhou, Jiangsu, China